CLINICAL TRIAL: NCT00397748
Title: PET Scanning of Brain Dopaminergic Signal Transduction Involving Arachidonic Acid in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: PET Scanning of Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060246; 06-M-0246
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2012-11-27

CONDITIONS: Volunteer; Attention Deficit Hyperactivity Disorder
Keywords: Phospholipase A2; D2 Receptors; Apomorphine; Trimethobenzamide; Attention Deficit Hyperactivity Disorder; ADHD; Healthy Volunteer; HV
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will explore the brain in men with and without attention deficit hyperactivity disorder (ADHD). It will use positron emission tomography (PET) and magnetic resonance imaging (MRI) to study brain function and nerve cell communication involving phospholipids (fatty molecules that make up the covering of nerve cell fibers in the brain and are involved in communication between the cells). It will also look at how nerve cell communication is related to blood flow. In particular, the study will explore communication through the dopamine system, which is one of the main neurotransmitter systems in the brain involved in ADHD.

Healthy men and men with ADHD between 18 and 55 years of age may be eligible for this study.

Participants undergo the following procedures:

"<TAB>Medical history and psychiatric and medical evaluation, including blood and urine tests.

"<TAB>MRI scan. This test uses a strong magnetic field and radio waves to obtain images of the brain. The subject lies still on a table that slides into the scanner (a metal cylinder) during the scanning.

"<TAB>PET scanning. The subject lies on the scanner bed with his head held still using a special facemask. A catheter (plastic tube or needle) is placed in an artery to collect blood samples and in a vein to inject radioactive isotopes for measuring blood flow and phospholipid metabolism. Scans are done after an injection of a saline solution and again after injection of apomorphine, a medication that turns on dopamine receptors in the brain. The injections are given under the skin of the abdomen, about one and a half hours apart....

DETAILED DESCRIPTION:
A. Objective

Attention deficit hyperactivity disorder (ADHD) is a heritable neurodevelopmental disorder with a reported male predominance that persists into adulthood and leads to significant morbidity in affected individuals. ADHD is currently hypothesized to reflect central dopaminergic dysfunction. Evaluation of human dopaminergic dysfunction using in vivo neuroimaging has been limited to studies of receptor localization and quantification, and dopamine synthesis, rather than direct measurement of the functional status of receptor signaling. There exists a need to thoroughly elucidate mechanisms underlying aberrant dopaminergic neurotransmission downstream of receptor activation in signaling processes. We have developed an in vivo method to measure neuroreceptor-initiated signal transduction involving activation of phospholipase A(2) to release the second messenger, arachidonic acid (AA). We propose to use positron emission tomography (PET) to quantitatively image dopamine-initiated signal transduction via AA in ADHD patients and healthy volunteers, in subjects administered the dopaminergic agonist, apomorphine, and to measure regional cerebral blood flow (rCBF) as well. We hypothesize that signaling and flow responses to apomorphine will be elevated, demonstrating hypersensitivity of the dopamine signaling mechanism.

B. Study population

18 healthy male volunteers between the ages of 18 and 55, will be recruited for this study (see justification for recruitment of males only in Study Design and Methods).

C. Design

All subjects will have up to four study-related visits to the Clinical Center in Bethesda over a one-year period, including an overnight stay. Participants will also be asked to complete an initial comprehensive telephone questionnaire to elicit whether they meet criteria for study participation, followed by on-site visits to NIH to complete a modified battery of neuropsychiatric screening tests related to symptom presence and severity. Questions relating to medical, family, psychiatric and developmental histories and lifestyle will be asked. In addition, visits will include a physical exam as well as blood and urine collection, and structural magnetic resonance imaging (MRI) of the head. Subject participation will culminate with sequential subcutaneous administration of a single dose of control vehicle solution (control) followed by the dopamine agonist apomorphine (after appropriate pre-medication with the anti-emetic, trimethobenzamide) or two sequential injections of vehicle for PET scans with attendant radiolabeled compounds.

D. Outcome Parameters

This study has four specific aims. First, regional cerebral blood flow will be quantified in response to an acute challenge with apomorphine s.c. and compared between study groups (ADHD/non-ADHD). Second, dopamine D(2)-like receptor signal transduction will be evaluated by PET in response to an acute challenge with apomorphine s.c. and compared between study groups (ADHD/non-ADHD). Third, baseline esterified and unesterified serum fatty acids will be compared between patients and control subjects. Lastly, we will examine the acute effect of apomorphine in the stimulation of serum growth hormone in all subjects, as confirmatory evidence for stimulation of central dopaminergic receptors.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must have normal values on screening measures to be in the study. They must be male and between 18 and 55 years of age. Primary efforts will also be to recruit non-smokers, given nicotine s ability to release dopamine presynaptically, a confound for this study. Previous smokers who have been abstinent for greater than 1 year may be considered.

EXCLUSION CRITERIA:

In addition to psychiatric criteria described above: past or current medical condition that would interfere with brain function - history of alcoholism, tobacco use (must have minimum of one year of full remission/complete abstinence from nicotine), neurological illness, head trauma with loss of consciousness, history of exposure to central nervous system toxin; history of central nervous system infection; metabolic, endocrine, connective tissue disease; hypertension or other cardiovascular disorder; gastrointestinal disorders; abnormal renal, liver or pulmonary function; blood dyscrasias; malignancy; nonstimulant or stimulant pharmacotherapy within 1 month of the study, or any history of antipsychotic medication; neurodegenerative or neurodevelopmental disorder; stroke; epilepsy; sensitivity to flashing lights; subjects requiring regular medication; subjects demonstrated by drug screening to have taken a controlled substance; subjects with a history of hypersensitivity to lidocaine; subjects with IQ less than 80. Females, adolescents and children will be excluded.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-09-15; Study Completion 2012-11-27

CONTACTS AND LOCATIONS:
Overall Officials: Judith L Rapoport, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Agid Y, Pollak P, Bonnet AM, Signoret JL, Lhermitte F. Bromocriptine associated with a peripheral dopamine blocking agent in treatment of Parkinson's disease. Lancet. 1979 Mar 17;1(8116):570-2. doi: 10.1016/s0140-6736(79)91003-1. PMID 85162
- [Background] Amenta F, Ricci A, Tayebati SK, Zaccheo D. The peripheral dopaminergic system: morphological analysis, functional and clinical applications. Ital J Anat Embryol. 2002 Jul-Sep;107(3):145-67. PMID 12437142
- [Background] Axelrod J. Phospholipase A2 and G proteins. Trends Neurosci. 1995 Feb;18(2):64-5. doi: 10.1016/0166-2236(95)93873-v. No abstract available. PMID 7537411